CLINICAL TRIAL: NCT01615640
Title: Monitoring the Response of Osteosarcoma Under Neoadjuvant Chemotherapy: The Value of Dynamic Contrast Enhancement and Diffusion-weighted MRI
Brief Title: Diffusion Study on Patients With Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Klinikum Stuttgart (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Dr. Thekla von Kalle, Dr. Thekla von Kalle, Klinikum Stuttgart
Other Study IDs: 02.08.2010 V.1.0
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Response of chemotherapy; Dynamic contrast medium examination; Diffusion-weighted MR imaging
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteosarcoma patients: Patients with an histologically proven osteosarcoma will be entered into the study.

SUMMARY:
The aim of the study is to assess the accuracy of dynamic contrast enhanced and diffusion-weighted MR Imaging in evaluating response to chemotherapy in osteosarcoma.

DETAILED DESCRIPTION:
Dynamic contrast-enhanced and diffusion-weighted magnetic resonance imaging have the potential to measure early cellular and vascular changes that occur in response to chemotherapy and could therefore be early predictors of therapeutic response.

Aim of our study is to assess the accuracy of dynamic contrast enhanced and diffusion-weighted MR imaging in evaluating response to chemotherapy during the preoperative treatment of osteosarcoma. Patients will undergo dynamic contrast-enhanced and diffusion-weighted magnetic resonance imaging before, during and after chemotherapy.

Our long-term goal is to use these imaging techniques to develop non-invasive methodologies that would be better predictors of tumor response than the current clinical standard and earlier predictors than histological evaluation of the whole tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of osteosarcoma of all entities
* Written informed consent of patient

Exclusion Criteria:

* No written informed consent
* Contraindications to MRI (pacemaker, aneurysm clip, mechanical and/or electrical device or metallic fragment, severe claustrophobia)
* Severe, active co-morbidity
* Major medical illnesses or psychiatric impairments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: German, Austrian and Swiss patients with an osteosarcoma will be entered into the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thekla von Kalle, Doctor, Principal Investigator — Klinikum Stuttgart
Locations (1):
- Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg, Germany